CLINICAL TRIAL: NCT01438008
Title: Be Sweet to Sick Babies: Analgesic Effects of Oral Sucrose and Concomitant Opioid Analgesics; a Pilot Randomized Controlled Trial
Brief Title: Pilot Study of Sucrose to Reduce Pain in Sick Babies
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Feasibility of study at single site; changes in clinical practice in opioid use
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Denise Harrison, Endowed Chair in Nursing Care of Children, Youth and Families, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 123942
Record Dates: First submitted 2011-09-16; First posted 2011-09-21 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Pain Due to Certain Specified Procedures
Keywords: Sucrose; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucrose 24% po (Experimental): 24% sucrose solution. The Children's Hospital of Eastern Ontario (CHOE) pharmacy department will provide syringes labeled "NICU Pain Relief Study" containing a maximum dose of 1 mL of a 24% sucrose solution
  Interventions: Drug: 24% sucrose po solution
- Placebo po (Placebo Comparator): The CHEO pharmacy department will provide a syringe labeled "NICU Pain Relief Study" containing a maximum of 1 ml dose of water (contents almost identical in color, consistency and odor to the sucrose solution) in identical packagings
  Interventions: Drug: Placebo po

INTERVENTIONS:
Drug: 24% sucrose po solution — CHEO pharmacy department will provide syringes labeled "NICU Pain Relief Study" containing a maximum of 1 ml dose of a 24% sucrose solution. The maximum amount of the study solution will be administered according to the infant's gestational age and according to the hospital's Sucrose policy. The total amount of the study solution will be divided into a maximum of 5 aliquots and administered throughout the procedure at two minutes prior to the heel lance, immediately prior to the heel lance, and two-minutely intervals until completion of the procedure.
  Other Names: CHEO Sucrose
  Arms: Sucrose 24% po
Drug: Placebo po — CHEO pharmacy department will provide syringes labeled "NICU Pain Relief Study" containing a maximum of 1 ml dose of water (almost identical in color, consistency and odor placebo to the sucrose solution in identical packaging) The total amount of the study solution will be divided into 5 aliquots and administered throughout the procedure at two minutes prior to the heel lance, immediately prior to the heel lance, and two-minutely intervals until completion of the procedure
  Other Names: Baxter sterile water
  Arms: Placebo po

SUMMARY:
Small amounts of sweet tasting sugar water reduces pain in babies during painful blood tests and injections. The investigators do not know if sugar also reduces pain in babies already receiving a continuous infusion of opioid analgesics. This project will help determine if small amounts of sugar water reduce pain in babies already receiving a continuous infusion of opioid analgesic during a heel lance procedure or nasogastric/orogastric (NG/OG) tube insertions. The investigators hypothesize that infants who are receiving opioid analgesics will have lower pain scores during their blood tests (heel lance) or NG/OG tube insertion, when sucrose is given, compared to when water is given.

DETAILED DESCRIPTION:
Background: Sick infants nursed in Neonatal Intensive Care Units (NICU) are exposed to large numbers of repeated painful procedures during their hospitalization [1-6]. Effectively reducing pain during these frequently performed and repeated painful procedures minimizes short term behavioural and physiological responses to pain, and has the potential to reduce long term adverse effects, including altered responses to subsequent pain [7] and increased risk of adverse neurodevelopmental, behavioural, and cognitive outcomes [8] The effectiveness of sucrose and other sweet solutions in the reduction of pain during painful procedures in infants has been well established. Despite the large numbers of randomized controlled trials (RCTs) of sweet solutions for procedural pain reduction in infants, there remain significant knowledge and research gaps. One of the key unanswered questions is whether sweet solutions reduce pain when given with concomitant opioid analgesics [9].

Rationale: Sick infants in hospital need to have blood tests as part of their medical care. Oral sucrose and glucose has shown to effectively reduce behavioural responses to pain and pain scores during commonly performed painful procedures in preterm and term newborn infants and infants up to 12 months of age. However, the investigators do not know if this also works for infants already receiving a continuous infusion of opioid analgesics. The aim is to establish preliminary evidence of the effectiveness of oral sucrose in reducing pain during heel lancing or NG/OG tube insertion when concomitant opioid analgesics are being administered, and to use the pilot data to inform a full scale RCT.

Hypothesis: Infants who are receiving opioid analgesics will have lower pain scores during their blood tests (heel lance) or NG/OG tube insertion, when sucrose is given, compared to when water is given.

Primary Objective: To obtain preliminary data about the effectiveness of sucrose and concomitant opioid analgesics compared to opioid analgesics alone during the painful procedure of heel lancing or NG/OG tube insertion to inform a full scale RCT.

Secondary Objectives: To determine the acceptability of the interventions to infants' parents and to use these results to help us calculate sample size for a subsequent full trial.

Methods: A single-center, randomized, double-blind, placebo controlled pilot trial will be conducted in an urban tertiary care pediatric university-affiliated hospital NICU. The study population is all infants who are inpatients in the Neonatal Intensive Care Unit (NICU) who are receiving a continuous infusion of opioid analgesics and who require a heel lance for the purpose of medically-required capillary blood sampling or a NG/OG tube insertion. Study participants will be randomly allocated to receive 24% sucrose solution or a placebo solution (water). The maximum amount of the study solution will be administered according to the infant's gestational age and according to the hospital's Sucrose policy:

<28 weeks gestation = maximum dose of 0.1 mL; 28-31 weeks gestation = maximum dose of 0.3 mL; 32-35 weeks gestation = maximum dose of 0.5 mL; >36 weeks gestation = maximum dose between 0.5-1.0 mL.

The primary outcome measure is the difference in pain levels during the heel lance procedure or NG/OG tube insertion in the study population as assessed by the Premature Infant Pain Profile (PIPP).

Secondary outcomes will include; i) total crying time; ii) skin conductance activity, a valid, non-invasive, physiological measure of pain and stress in infants.

Statistical analysis: PIPP scores, crying time, and skin conductance activity will be summarized using mean and standard deviation if normally distributed, and median and interquartile range (IQR) if non-normally distributed. An intention to treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

Infants who are inpatients of the NICU:

* Who are receiving a continuous intravenous infusion of an opioid analgesic such as morphine or fentanyl at a maximum dose equivalent to 20 mcg/kg/hr of morphine and;
* Who require heel lance for medically required blood sampling or nasogastric/orogastric (NG/OG) tube insertions and;
* Who are eligible to receive sucrose as per the hospital's Sucrose policy for infants.

Exclusion Criteria:

* Infants less than 25 weeks gestation
* Infants with any injury to the skin where the probe needs to be placed
* Infants with an implanted defibrillator or pacemaker
* Infants with an injury affecting sympathetic nerve conduction
* Infants exposed to antenatal methadone
* Infants who, aside from being on opioid analgesics, are ineligible to receive sucrose as per the hospital's Sucrose policy38
* If the infant's mother wishes to breastfeed during the procedure
* Infants with known or suspected fructose intolerance
* Infants with spinal cord malformation (e.g. myelomeningocele and sacral teratoma) since these infant's response, and sensitivity to pain may differ from infants without spinal cord malformations
* Infants who are unconscious, heavily sedated and those with absent gag and/or swallow reflex
* Infants who are in isolation with only essential personnel caring for them
* To ensure there is no interaction effect of muscle relaxants, which may impact on infants' ability to mount a behavioural response to pain, assessments will not be conducted until a period of 24 hours since the previous muscle relaxant dose
* Parental language barrier (if unable to speak/understand French and/or English)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Harrison, PhD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Barker DP, Rutter N. Exposure to invasive procedures in neonatal intensive care unit admissions. Arch Dis Child Fetal Neonatal Ed. 1995 Jan;72(1):F47-8. doi: 10.1136/fn.72.1.f47. PMID 7743285
- [Background] Carbajal R, Rousset A, Danan C, Coquery S, Nolent P, Ducrocq S, Saizou C, Lapillonne A, Granier M, Durand P, Lenclen R, Coursol A, Hubert P, de Saint Blanquat L, Boelle PY, Annequin D, Cimerman P, Anand KJ, Breart G. Epidemiology and treatment of painful procedures in neonates in intensive care units. JAMA. 2008 Jul 2;300(1):60-70. doi: 10.1001/jama.300.1.60. PMID 18594041
- [Background] Harrison D, Loughnan P, Manias E, Johnston L. Analgesics administered during minor painful procedures in a cohort of hospitalized infants: a prospective clinical audit. J Pain. 2009 Jul;10(7):715-22. doi: 10.1016/j.jpain.2008.12.011. Epub 2009 Apr 23. PMID 19398379
- [Background] Johnston CC, Collinge JM, Henderson SJ, Anand KJ. A cross-sectional survey of pain and pharmacological analgesia in Canadian neonatal intensive care units. Clin J Pain. 1997 Dec;13(4):308-12. doi: 10.1097/00002508-199712000-00008. PMID 9430811
- [Background] Porter FL, Anand KJ. Epidemiology of Pain in Neonates. Research & Clinical Forums 20(4): 9-16, 1998.
- [Background] Simons SH, van Dijk M, Anand KS, Roofthooft D, van Lingen RA, Tibboel D. Do we still hurt newborn babies? A prospective study of procedural pain and analgesia in neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1058-64. doi: 10.1001/archpedi.157.11.1058. PMID 14609893
- [Background] Taddio A, Katz J. The effects of early pain experience in neonates on pain responses in infancy and childhood. Paediatr Drugs. 2005;7(4):245-57. doi: 10.2165/00148581-200507040-00004. PMID 16117561
- [Background] Grunau RE, Holsti L, Haley DW, Oberlander T, Weinberg J, Solimano A, Whitfield MF, Fitzgerald C, Yu W. Neonatal procedural pain exposure predicts lower cortisol and behavioral reactivity in preterm infants in the NICU. Pain. 2005 Feb;113(3):293-300. doi: 10.1016/j.pain.2004.10.020. PMID 15661436
- [Background] Harrison D, Loughnan P, Manias E, Smith K, Johnston L. Effect of concomitant opioid analgesics and oral sucrose during heel lancing. Early Hum Dev. 2011 Feb;87(2):147-9. doi: 10.1016/j.earlhumdev.2010.11.008. Epub 2010 Dec 8. PMID 21138786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2012 and September 2015, 73 infants admitted in the NICU were assessed for eligibility, 50 (69%) were ineligible, of the 23 (32%) infants that were approached, 7 (3%) declined to participate, 16 (70%) provided consent.
Pre-assignment Details: Consent was obtain for 16 infants to participate, 7 (44%) were not randomized (prior to data collection n=3 infants were weaned off fentanyl, n=3 infants were discharged/transferred, n=1 medical team refused). 9 (12%) infants were randomized. 4 infants were allocated to sucrose and 5 infants were allocated to water.
Groups:
- Sucrose 24% po: 24% sucrose solution. The CHEO pharmacy department will provide syringes labeled "NICU Pain Relief Study" containing a maximum dose of 1 mL of a 24% sucrose solution
  24% sucrose po solution: CHEO pharmacy department will provide syringes labeled "NICU Pain Relief Study" containing a maximum of 1 ml dose of a 24% sucrose solution. The maximum amount of the study solution will be administered according to the infant's gestational age and according to the hospital's Sucrose policy. The total amount of the study solution will be divided into a maximum of 5 aliquots and administered throughout the procedure at two minutes prior to the heel lance, immediately prior to the heel lance, and two-minutely intervals until completion of the procedure.
Period: Overall Study
Arm/Group | Sucrose 24% po | Placebo po
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sucrose 24% po | Placebo po | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 17.5 [5 to 36] | 10.0 [6 to 67.5] | 10.0 [5 to 42.5]
Age, Continuous [Median (Inter-Quartile Range); unit: gestational age (days)] | 261.5 [206.75 to 289.25] | 236.0 [177 to 265.5] | 236.0 [187.5 to 278]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 3 | 4
Type of Procedure [Count of Participants; unit: Participants]
  Heel lance | 4 | 4 | 8
  Naso/oro gastric insertion | 0 | 1 | 1
Duration of Procedure [Median (Inter-Quartile Range); unit: seconds] | 281 [137 to 344.75] | 380 [182 to 494] | 301 [179 to 385]
Type of opioid administered [Count of Participants; unit: Participants]
  Morphine | 1 | 1 | 2
  Fentanyl | 3 | 4 | 7
Previous use of sucrose [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 1 | 1 | 2
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Premature Infant Pain Profile (PIPP)
Description: The Premature Infant Pain Profile (PIPP), a validated seven-indicator multidimensional pain assessment tool which is extensively used in neonatal pain research. The scale consists of seven indicators including assessment of gestational age and behavioural state (contextual indicators), heart rate and oxygen saturation (physiological indicators), and facial actions-brow bulge, eye squeeze, and nasolabial furrow (behavioural indicators), which are scored on a 0-3 scale and added for a total score of 0-21 Facial expression scores were also recorded on a 0-4 scale using a modified Neonatal Facial Coding System (NFCS) at 30, and 60 seconds following the beginning of the procedure. The modified NFCS coded for the presence (1) or absence (0) of the 4 most common facial expressions in response to acute pain (brow bulge, eye squeeze, nasolabial furrow, and stretch open mouth).
  High values on both of these scales represent worse outcome (i.e higher pain intensity).
Time Frame: Baseline, day one of blood test
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sucrose 24% po | Placebo po
Number analyzed (Participants) | 4 | 5
score on a scale
  PIPP-R at 30 seconds | 9.5 [7.5 to 13.75] | 10 [3.5 to 11.5]
  PIPP-R at 60 seconds | 9.5 [6.25 to 14.25] | 9 [4 to 14]
  NFCS at 30 seconds | 1.5 [0.25 to 3.5] | 0 [0 to 3]
  NFCS at 60 seconds | 2 [0 to 4] | 0 [0 to 3]

2. Secondary Outcome: Total Crying Time
Description: Cry duration is a useful method to determine infant distress in general and to evaluate pain in the infant's environmental context.
Time Frame: Total crying time were recorded as a proportion of the time spent crying over the total length of procedure and/or in the 3 minutes that followed.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Sucrose 24% po | Placebo po
Number analyzed (Participants) | 4 | 5
seconds | 0 [0 to 147.1275] | 0 [0 to 102.685]

ADVERSE EVENTS:
Arm/Group | Sucrose 24% po | Placebo po
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Recruitment for this study was difficult due to the tight inclusion criteria. Although consent was provided for 16 infants to participate, only 9 infants were randomized and studied the results may contribute to systematic review data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No